CLINICAL TRIAL: NCT00004046
Title: A Phase II Study of Intravenous DX-8951f Administered Daily for Five Days Every Three Weeks to Patients With Metastatic Adenocarcinoma of the Breast
Brief Title: Chemotherapy in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067148; DAIICHI-8951A-PRT011; MDA-ID-98308
Record Dates: First submitted 2000-05-02; First posted 2004-04-15 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DX-8951f in treating women who have metastatic breast cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of DX-8951f in women with metastatic adenocarcinoma of the breast who have failed prior therapy with an anthracycline and a taxane. II. Evaluate the quantitative and qualitative toxicities of this drug in these patients. III. Evaluate the pharmacokinetics of this drug in these patients.

OUTLINE: Patients receive DX-8951f IV over 30 minutes daily for 5 days. Courses repeat every 21 days. Treatment continues in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic adenocarcinoma of the breast Prior treatment with an anthracycline (e.g., doxorubicin or epirubicin) and a taxane (e.g., paclitaxel or docetaxel) either as adjuvant therapy or for advanced disease Bidimensionally measurable disease Sentinel lesions must be outside of any prior radiation port No resected disease or stage IV with no evaluable disease No brain metastases or leptomeningeal disease No symptomatic lymphangitic pulmonary metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Hemoglobin at least 9.0 g/dL Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT or SGPT no greater than 2 times upper limit of normal (ULN) (5 times ULN if liver metastases present) Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No active congestive heart failure No uncontrolled angina No myocardial infarction within past 6 months Neurologic: No history of an existing grade 3-4 peripheral neuropathy of any etiology Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No allergy to camptothecin or its derivatives No concurrent serious infection No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix No overt psychosis, mental disability, or incompetence No other life threatening disease

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy No prophylactic colony stimulating factors to prevent neutropenia (except when neutropenia fever occurs despite dose reduction) Chemotherapy: See Disease Characteristics No greater than 3 prior chemotherapy regimens for metastatic breast cancer or as either adjuvant or neoadjuvant therapy At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered No other concurrent cytotoxic chemotherapy Endocrine therapy: Exogenous hormonal therapy for stage IV disease and/or as adjuvant therapy allowed At least 3 weeks since prior hormonal therapy except for: Patients who are highly unlikely to have a withdrawal response to cessation of hormonal therapy (e.g., patients with disease that is primarily resistant to hormonal therapy, patients without prior partial response, or stabilization of disease lasting less than 6 months) Patients with new or extensive visceral metastases Patients with rapidly progressive or symptomatic metastases during hormonal therapy Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No prior radiotherapy to greater than 50% of bone marrow No concurrent radiotherapy Surgery: See Disease Characteristics At least 4 weeks since prior major surgery and recovered No concurrent surgery Other: No other concurrent anticancer treatment At least 28 days since other prior investigational drugs, including analgesics or antiemetics No other investigational drugs during and for 28 days after the study No drugs that induce or inhibit CYP3A enzyme

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States